CLINICAL TRIAL: NCT00235053
Title: A Pilot Study to Assess the Incidence of Local Oropharyngeal and Laryngeal Adverse Effects of Advair DISKUS 250/50 mcg BID as Assessed by the Development of Laryngitis and Oropharyngeal Candidiasis in Adults With Mild Persistent Asthma
Brief Title: Study to Assess the Incidence of Local Oropharyngeal and Laryngeal Adverse Effects of Advair DISKUS 250/50 mcg BID
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergy & Asthma Medical Group & Research Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NONE0-L00081
Record Dates: First submitted 2005-10-06; First posted 2005-10-10 (Estimated); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Asthma; Candidiasis, Oral; Voice Disorders
Keywords: asthma; candidiasis, oral; voice disorders
MeSH Terms: conditions — Asthma; Candidiasis, Oral; Voice Disorders | interventions — Fluticasone

INTERVENTIONS:
Drug: fluticasone/salmeterol DISKUS 250/50

SUMMARY:
This Pilot study is designed to explore the rate of local side effects of fluticasone as delivered by Advair and to determine the best outcome measure to assess these effects. This study is the initial step, and will be followed by a larger scale study.

DETAILED DESCRIPTION:
Asthma is a chronic inflammatory disorder of the airways. The inflammation is associated with bronchial hyperresponsiveness, airflow obstruction, and respiratory symptoms including wheezing, coughing and chest tightness.

Inhaled corticosteroids are the most effective controller asthma medications. They are indicated for management of persistent asthma at all levels of severity. They have been documented to improve symptoms and pulmonary function and reduce exacerbations, need for quick-relief medications and airway hyperresponsiveness.

Despite their benefits, inhaled corticosteroids have been associated with adverse local effects. These include oral candidiasis and dysphonia. However, though these risks have been reported, they have not been carefully studied. The incidence of oral candidiasis in newly treated subjects and its onset within a carefully monitored timeframe have not been adequately assessed.

A more overtly undesirable effect is dysphonia. Data on it are usually collected from spontaneous reports by patients in clinical trials. However, awareness of dysphonia requires a certain degree of subjective discomfort to initiate the report. Subjective awareness of dysphonia often varies based on an individuals voice requirements. A singer, for example, is usually acutely aware of minor voice changes in contrast to someone who does not depend on voice quality. Nonetheless, voice abnormalities can probably occur with similar frequency in patients who are concerned or not concerned with their voice due to inhaled corticosteroids. New subjective scales for reporting on an individual's voice have recently been validated and published in other areas. These scales have not been validated in patients with asthma or in subjects using inhaled corticosteroids. New technologies for objective voice assessment have also been developed and these permit greater ability to quantify voice changes. These advances permit better measures of the potential adverse effects of inhaled corticosteroids on voice both with regard to onset of abnormalities and with regard to magnitude of effects.

This pilot study is an initial probe into clarifying the potential of the inhaled corticosteroid, fluticasone propionate delivered in the Advair DISKUS device to produce oral candidiasis and voice changes, and to determine the best measurement to quantitate objectively that effect.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female, 18-55 years of age. Females will be eligible only if they are:

   1. Surgically sterilized, post-menopausal, abstinent, or practicing adequate method of birth control, and if they have a
   2. Negative urine pregnancy test (females of childbearing potential)
2. History of mild persistent asthma for at least 6 months as defined by NIH NHLBI April 19971

At Visit 1 (Screening) treatment for the last 30 days prior to screening must be:

* No inhaled corticosteroid therapy. (Previous use of leukotriene receptor antagonists, and/or cromones, in addition to bronchodilators also allowed.)

Exclusion Criteria:

1. Female subjects who are pregnant or trying to become pregnant
2. Breast feeding
3. Current patient reported hoarseness or sore throat
4. Presence of oropharyngeal thrush (as determined by investigator examination without culture results)
5. Unresolved fungal, viral or bacterial infection elsewhere in the body
6. Viral or bacterial respiratory tract infection within the last 14 days
7. History of persistent gastro-esophageal reflux refractory to conventional treatment within the last 30 days
8. Has smoked within the previous 6 months or has greater than a lifetime 10 pack-year smoking history or regular exposure to environmental tobacco smoke
9. History of inflammatory arthritis requiring immunosuppressive or corticosteroid therapy
10. History of glaucoma, cataracts (lens opacities), retinal disease, or blindness
11. Any serious concomitant disease such as cancer or serious renal, hepatic, cardiac, immunodeficiency, neurological, psychiatric, or other disease
12. Any medical condition that, in the judgment of the investigator, might interfere with the study, require treatment or make implementation of the protocol or interpretation of the study results difficult
13. Active or quiescent tuberculosis infections of the respiratory tract
14. History of chronic bronchitis, COPD or emphysema
15. History of alcohol abuse (more than 2 drinks/day on average) or drug abuse within the past 2 years
16. History within the last 2 years of moderate asthma requiring prednisone on more than two occasions per year
17. Treatment with any investigational drug within the past 30 days
18. More than 1 short (less than 2 weeks) course of systemic corticosteroids in the previous year prior to screening (Visit 1) or have had systemic corticosteroids in the past pervious 2 months prior to Visit 1.
19. Subjects can be on maintenance immunotherapy but cannot have begun an immunotherapy regimen or have had a change in their immunotherapy regimen within 30 days prior to screening (Visit 1).
20. Subjects may be on intranasal steroid if it has been maintained for 4 weeks prior to screen and a constant stable dose is maintained for the duration of the trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13
Dates: Start 2005-08; Study Completion 2005-11

PRIMARY OUTCOMES:
To determine the magnitude of change from baseline to end of study in the Voice Handicap Index (VHI) with Advair® DISKUS 250/50 mcg BID in subjects with mild persistent asthma.

SECONDARY OUTCOMES:
1. Voice Related Quality of Life (VRQOL)
2. Inhaled Corticosteroid Questionnaire (ICQ)
3. Reflux Symptom Index (RSI)
4. Videostroboscopy and Determination of Reflux Finding Score (RFS)
5. Voice jitter
6. Voice shimmer
7. Signal to noise ratio
8. Oropharyngeal Candida species culture
9. Oropharyngeal Candida species related symptoms
10. Oropharyngeal thrush on physical exam

CONTACTS AND LOCATIONS:
Overall Officials: Eli O Meltzer, MD, Principal Investigator — Allergy & Asthma Medical Group & Research Center
Locations (1):
- Allergy & Asthma Medical Group & Research Center, San Diego, California, United States